CLINICAL TRIAL: NCT00753038
Title: Phase 2 Study of Intravenous Administration of a Wild-Type Reovirus (REOLYSIN®) in Combination With Paclitaxel and Carboplatin in Patients With Platinum-Refractory Metastatic and/or Recurrent Squamous Cell Carcinoma of the Head and Neck.
Brief Title: Phase 2 Study of REOLYSIN® in Combination With Paclitaxel and Carboplatin in Patients With Head and Neck Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oncolytics Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REO 015
Record Dates: First submitted 2008-09-12; First posted 2008-09-16 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Carcinoma, Squamous Cell of the Head and Neck
Keywords: carcinoma; squamous cell; head; neck; REOLYSIN; chemotherapy; Carboplatin; Paclitaxel
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma | interventions — reolysin; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: REOLYSIN® — 3E10 TCID50, 1 hour intravenous infusion, administered on Days 1, 2, 3, 4 and 5 of a 21 day cycle
Drug: Carboplatin — 5 AUC mg/mL min, 30 min intravenous infusion, given on Day 1 of a 21 day cycle
Drug: Paclitaxel — 175 mg/m2, 3 hour intravenous infusion, given on Day 1 of a 21 day cycle

SUMMARY:
The purpose of this Phase 2 study is to investigate whether intravenous administration of REOLYSIN® therapeutic reovirus in combination with Paclitaxel and Carboplatin is effective and safe in the treatment of squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
Squamous cell carcinoma of the head and neck is the sixth most common cancer in the world. More than 50% of patients diagnosed with advanced regional disease will relapse locally or at distant sites. Initial therapeutic options include irradiation, surgery and chemotherapy. The most commonly used agents are cisplatin and carboplatin, generally in combination with 5-FU or a taxane. Erbitux has recently been approved for use in first-line with radiation and in second-line as monotherapy. Only about a third of the patients will respond to first-line platinum-based therapy and the median overall survival is 6-9 months.

Preliminary assessment of a Phase 1 study being conducted in the UK investigating the combination of REOLYSIN®, carboplatin and paclitaxel suggested that patients with head and neck carcinomas may represent a group of patients in whom this treatment combination is active.

This Phase 2 study is designed to characterize the efficacy and safety of REOLYSIN® given intravenously in combination with paclitaxel and carboplatin every 3 weeks in patients with squamous cell carcinoma of the head and neck.

Response is a primary endpoint of this trial. Patients will be clinically evaluated after each course of treatment and radiologically every other cycle. A complete or partial response must be confirmed at least 4 weeks after the first assessment that documents such a response and every two cycles thereafter.

The safety of the paclitaxel, carboplatin and REOLYSIN® combination will be assessed by the evaluation of the type, frequency and severity of adverse events, changes in clinical laboratory tests, immunogenicity and physical examination.

Patients may continue to receive therapy under this protocol, provided they have not experienced either progressive disease or unacceptable drug-related toxicity that does not respond to either supportive care or dose reduction.

ELIGIBILITY:
Inclusion Criteria:

* have platinum-refractory metastatic and/or recurrent histologically confirmed stage III/IV squamous cell carcinoma of the head and neck (oral cavity, larynx or pharynx) with no secondary cancers
* have evidence of measurable disease
* have documented progressive disease (PD) on or within 190 days following the completion of treatment of cisplatin-based or carboplatin-based chemotherapy in a recurrent or metastatic setting and if treatment with cetuximab was considered indicated for the patient, documented PD(on or within 190 days of treatment)
* have no continuing acute toxic effect of any prior radiotherapy, chemotherapy or surgical procedures
* have received no chemotherapy, radiotherapy, immunotherapy or hormonotherapy within 28 days
* have ECOG performance score of ≤2
* have life expectancy of at least 3 months
* absolute neutrophils ≥ 1.5 x10^9/L; platelets ≥100 x10^9; hemoglobin ≥9.0 g/dL; serum creatinine ≤1.5 xULN; bilirubin ≤1.5 x ULN; AST/ALT ≤2.5xULN
* negative pregnancy test for females of childbearing potential

Exclusion Criteria:

* have known brain metastasis
* have known bone metastasis
* be on immunosuppressive therapy; have known HIV infection or active hepatitis B or C
* be a pregnant or breast-feeding woman
* have clinically significant cardiac disease
* have dementia or altered mental status that would prohibit informed consent
* have any other severe, acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgement of the Principal Investigator, would make the patient inappropriate for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-08; Primary Completion 2011-07 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Determine the objective response rate (complete response (CR) + partial response (PR)) of the treatment regimen in the study population | For PR or CR, changes in tumor measurements must be confirmed 4 weeks after the criteria for response are first met.

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of the treatment regimen in the study population. | Within 30 days of last dose of REOLYSIN®
Determine the disease control rate (CR, PR and stable disease (SD)), duration of response, time to disease progression and survival with the treatment regimen in the study population. | For PR or CR, changes in tumor measurements must be confirmed 4 weeks after the criteria for response are first met. For SD, follow-up measurements must have met the SD criteria at least once after trial entry at a minimum interval of 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Mita, MD, Principal Investigator — Cancer Therapy and Research Center, Texas
Locations (2):
- United States (2):
  - Montefiore Medical Center, The Bronx, New York
  - Cancer Therapy and Research Center at UTHSCSA, San Antonio, Texas